CLINICAL TRIAL: NCT01965002
Title: A Feasibility Study to Evaluate the Safety and Effectiveness of ExAblate Magnetic Resonance Imaging Guided High Intensity Focused Ultrasound Treatment of Soft Tissue Tumors of the Extremities
Brief Title: Feasibility of ExAblate MRI Guided High Intensity Focused Ultrasound Tx of Soft Tissue Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Accrual factor
Sponsor: Pejman Ghanouni (Other)
Responsible Party: Sponsor-Investigator, Pejman Ghanouni, Assistant Professor of Radiology, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-26667; VAR0095 (Other: OnCore)
Record Dates: First submitted 2013-10-15; First posted 2013-10-17 (Estimated); Results first posted 2018-05-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-04

CONDITIONS: Soft Tissue Neoplasms
MeSH Terms: conditions — Soft Tissue Neoplasms | interventions — Aspirin; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (1):
- MRgHIFU (Experimental): The InSightec ExAblate 2000 magnetic resonance-guided high-intensity focused ultrasound (MRgHIFU) system is a non-invasive device that is fully integrated with an MR imaging system and used for the ablation of soft tissue. The treatment process begins with the physician acquiring a set of MR images, identifying 1+ target volume(s) of fibroid tissue to be ablated, and drawing the treatment contours. The therapy planning software computes the type and number of sonications required to treat the defined volume while minimizing total treatment time. MR images taken during the sonication provide a diagnostic quality image of the target tissue and a quantitative, real-time temperature map overlay to confirm the therapeutic effect of the treatment. The transducer is then automatically moved to the succeeding treatment point and the process is repeated until the entire volume has been treated. About 100 individual sonications can be delivered over a 3-hour period to complete a treatment.
  Interventions: Device: MRgHIFU; Drug: Aspirin; Drug: Enoxaparin

INTERVENTIONS:
Device: MRgHIFU — The InSightec ExAblate 2000 magnetic resonance-guided high-intensity focused ultrasound (MRgHIFU) system is a non-invasive thermal ablation device fully integrated with an MR imaging system and used for the ablation of soft tissue
  Other Names: ExAblate Magnetic Resonance Imaging Guided High Intensity Focused Ultrasound
Drug: Aspirin — 325 mg PO for deep venous thrombosis (DVT) prophylaxis initiated 2 hours prior to magnetic resonance-guided high-intensity focused ultrasound (MRgHIFU) treatment
  Other Names: Ecotrin
Drug: Enoxaparin — 40 mg by subcutaneous (SC) administration, for deep venous thrombosis (DVT) prophylaxis initiated 2 hours prior to magnetic resonance-guided high-intensity focused ultrasound (MRgHIFU) treatment
  Other Names: Lovenox

SUMMARY:
The goal of this project is to evaluate the safety and preliminary efficacy of ExAblate magnetic resonance-guided high-intensity focused ultrasound (MRgHIFU) surgery in the treatment of soft tissue tumors of the extremities.

DETAILED DESCRIPTION:
Given that the incidence of cancer increases with age, the number of elderly patients diagnosed and treated for soft tissue sarcomas (STS) will increase. The dilemma is that surgeons and medical oncologists may be hesitant to treat elderly patients in a comparably intensive manner as is used in the treatment of younger patients; factors such as decreased performance status, significant comorbidities, and disease natural history may erode enthusiasm for aggressive STS resection. To this end, a less invasive way of treating soft tissue tumors would be helpful in younger patients to minimize morbidity and in the elderly to provide less aggressive treatment options. The InSightec ExAblate 2000 magnetic resonance-guided high-intensity focused ultrasound (MRgHIFU) system is a non-invasive thermal ablation device fully integrated with an MR imaging system and used for the ablation of soft tissue (5-10). The ExAblate combines a focused ultrasound surgery (FUS) delivery system and a conventional diagnostic 1.5 T or 3 T MRI scanner. It provides a real-time therapy planning algorithm, thermal dosimetry, and closed-loop therapy control.

ELIGIBILITY:
INCLUSION CRITERIA

* ≥ 10 years of age.
* Benign or malignant soft tissue tumors of the extremities, flanks, pelvis, or shoulders requiring surgical intervention.
* Tumor must not have been treated previously with radiation.
* Targeted tumor(s) are accessible to the ExAblate device
* Targeted volume within the tumor is located deeper than 1 cm from the skin
* Targeted tumor is clearly visible by non-contrast magnetic resonance imaging (MRI)
* Karnofsky Performance Status > 60
* Normal platelet count and coagulation profile
* Glomerular filtration rate > 60 mL/min
* Able to safely undergo MRI exam and receive mild sedation for the treatment.
* Able to tolerate being in the MRI scanner for the duration of the study.
* Able and willing to give consent (or consent + assent where applicable), and able to attend all study visits.

EXCLUSION CRITERIA

* Previous radiation treatment to the tumor.
* Currently receiving dialysis.
* Acute medical condition (eg, pneumonia, sepsis) expected to hinder completion of the study
* Unstable cardiac status including:

  * Unstable angina pectoris on medication
  * Patients with documented myocardial infarction within six months of protocol entry
  * Congestive heart failure requiring medication (other than diuretic)
  * Patients on anti-arrhythmic drugs
* Severe hypertension (diastolic BP > 100 on medication)
* Contraindication for MR imaging such as implanted metallic devices that are not MRI-safe, size limitations, etc
* Severe hematologic, neurologic, or other uncontrolled disease
* Known intolerance or allergy to medications used for sedation (midazolam), analgesia (fentanyl), and local and regional anesthesia (lidocaine, bupivacaine, and ropivacaine)
* Known intolerance or allergy to MR contrast agent (gadolinium chelates) including advanced kidney disease
* Pregnant and nursing
* Karnofsky Performance Score < 60
* Severe cerebrovascular disease [cardiovascular accident (CVA) within 6 months]
* Not able or not willing to tolerate the required prolonged stationary position during treatment (up to 5 hrs of total table time)
* Target volume in tumor is less than 1 cm from neurovascular bundles, major blood vessels, bowel, or bladder.
* Targeted tumors:

  * NOT visible by non-contrast MRI, OR
  * NOT accessible to ExAblate device
* Not a candidate for either regional anesthesia or mild sedation
* Not be participating in another trial testing other investigational agents or devices

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-05; Primary Completion 2015-03-24 (Actual); Study Completion 2015-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raffi Avedian, MD, Principal Investigator — Stanford University; Pejman Ghanouni, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MRgHIFU
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- MRgHIFU: The InSightec ExAblate 2000 MRgHIFU system is a non-invasive device that is fully integrated with an MR imaging system and used for the ablation of soft tissue. The treatment process begins with the physician acquiring a set of MR images, identifying one or more target volume(s) of fibroid tissue to be ablated, and drawing the treatment contours. The therapy planning software computes the type and number of sonications required to treat the defined volume while minimizing total treatment time. MR images taken during the sonication provide a diagnostic quality image of the target tissue and a quantitative, real-time temperature map overlay to confirm the therapeutic effect of the treatment. The transducer is then automatically moved to the succeeding treatment point and the process is repeated until the entire volume has been treated. Approximately 100 individual sonications can be delivered over a 3-hour period to complete a treatment.
Arm/Group | MRgHIFU
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Safety - Incidence of Any Device-related Adverse Events
Description: Safety determined by evaluating for the incidence of any device-related adverse events. Patients will be assessed for pain and limb function, and by clinical examination before and after treatment to collect adverse events related to the treatment. Safety is reported as the total incidence of device-related adverse events.
Time Frame: 1 week
Population: All participants were evaluated for adverse events.
Measure: Number; unit: device-related adverse events
Groups:
- MRgHIFU: The InSightec ExAblate 2000 MRgHIFU system is a non-invasive thermal ablation device fully integrated with an MR imaging system being used for the ablation of tumor tissue
Arm/Group | MRgHIFU
Number analyzed (Participants) | 5
device-related adverse events | 8

2. Secondary Outcome: Adverse Event Severity
Description: Safety is further assessed by an evaluation of severity for the treatment-related adverse events, reported as the number of adverse events for each of the Common Terminology Criteria for Adverse Events (CTCAE) v4.0 grades.
  CTCAE Severity:
  1. mild
  2. moderate
  3. severe
  4. life-threatening
  5. fatal
Time Frame: 6 months
Measure: Number; unit: Treatment-related adverse events
Groups:
- MRgHIFU: In the resected tumor specimen, the volume of the ablated area will be determined by obtaining a digital photograph of each pathology slice. The region of interest corresponding to the ablated area will be traced, and the ablated area will be calculated for each slice and summed. Accuracy is assessed as the percent ablated volume relative to pre-treatment tumor volume.
Arm/Group | MRgHIFU
Number analyzed (Participants) | 5
Treatment-related adverse events
  CTCAE Grade 1 | 8
  CTCAE Grade 2 | 0
  CTCAE Grade 3 | 0
  CTCAE Grade 4 | 0
  CTCAE Grade 5 | 0

3. Secondary Outcome: Percent Successful Tumor Ablation
Description: In the resected tumor specimen, the volume of the ablated area will be determined by obtaining a digital photograph of each pathology slice. The region of interest corresponding to the ablated area will be traced, and the ablated area will be calculated for each slice and summed. Accuracy is assessed as the percent ablated volume relative to pre-treatment tumor volume.
Time Frame: Up to 1 week
Population: Due to the complexity of 3-dimensional mapping of tumors in soft tissues, the precision necessary to capture baseline tumor volume exceeded the capability of the equipment. Baseline data per protocol for the outcome calculation was only obtained from a single participant, resulting in an inability to conduct a robust per protocol analysis.
Measure: Number; unit: percent ablated volume
Arm/Group | MRgHIFU
Number analyzed (Participants) | 1
percent ablated volume | 40

ADVERSE EVENTS:
Time Frame: up to 10 months
Arm/Group | MRgHIFU
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MRgHIFU (N=5)
Pain at tumor site (General disorders) | 1 (1)
Edema at right distal thigh (Skin and subcutaneous tissue disorders) | 1 (1)
Mild backache from positioning (Musculoskeletal and connective tissue disorders) | 1 (1)
Diminished sensation along medial thigh (Musculoskeletal and connective tissue disorders) | 1 (1)
Mild erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Slight numbness along distal aspect of the incision (Musculoskeletal and connective tissue disorders) | 1 (1)
Mild pain at tumor site (Musculoskeletal and connective tissue disorders) | 1 (1)
Reduced range of motion in right knee (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No